CLINICAL TRIAL: NCT00002001
Title: The Antiviral Efficacy of Concurrent Zidovudine and 2',3'-Dideoxyinosine or 2',3'-Dideoxycytidine in Patients With Human Immunodeficiency Virus Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 052B; 02
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-09

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To evaluate the virologic effect of combined administration of zidovudine and ddI or ddC. To evaluate the immunologic effects of zidovudine and ddI or ddC. To evaluate combined administration of zidovudine and ddI or ddC for clinical efficacy. To evaluate the safety and the tolerance of the coadministration of zidovudine and ddI or ddC.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Patients with PCP may be randomized to study medication after contacting the sponsor and following a minimum 7-day course of therapy resulting in stabilization of their disease. Patients with stabilized disease must have fever < 39 C for at least 48 hours, p02 (on room air) > or = 60 mm and an A/A gradient < or = 30 mm.
* Prophylaxis for PCP.

Patients must have the following:

* HIV-1 seropositive by any federally licensed ELISA.
* Willingness to give informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Any immediately life-threatening infection or medical condition present at time of study entry.
* Any active opportunistic infection requiring chronic therapy with any of the agents listed in the exclusion concurrent medication section.
* Neoplasms other than basal cell carcinoma or in situ carcinoma of the cervix.
* Kaposi's sarcoma with visceral involvement or requiring systemic cytotoxic chemotherapy.
* AIDS dementia complex, > or = Stage 2.
* History of zidovudine induced toxicity.
* Prior history of acute pancreatitis during the past two years or chronic pancreatitis.
* Grade 2 neuropathy.
* Intractable diarrhea.
* History of seizures within the past six months or current requirement of anticonvulsants.
* Past or current heart disease.
* Fever > 39 C at entry.

Concurrent Medication:

Current requirement of anticonvulsants.

* Excluded:
* It is intended that patients developing new opportunistic infections during the course of the study will continue study participation, unless required therapy is associated with significant neurologic or hematologic toxicities, in which case the study medication may be temporarily discontinued.
* Ganciclovir.
* Chloramphenicol.
* Cisplatinum.
* Iodoquinol.
* Systemic Pentamidine.
* Disulfiram.
* Ethionamide.
* Glutethimide.
* Gold.
* Hydralazine.
* Metronidazole.
* Sodium Cyanate.
* Thalidomide.
* Vincristine.
* Allopurinol.
* Probenecid.

Concurrent Treatment:

Excluded:

* Radiation therapy. (with the exception of electron beam therapy to an area of < 100cm/m2.)

Patients with the following are excluded:

* Any immediately life-threatening infection or medical condition present at time of study entry.
* Any active opportunistic infection requiring chronic therapy with any of the agents listed in the exclusion concurrent medication section.
* Active alcohol or drug abuse, sufficient in the investigator's opinion to prevent compliance with study therapy.
* Neoplasms other than basal cell carcinoma or in situ carcinoma of the cervix.
* Kaposi's syndrome with visceral involvement or requiring systemic cytotoxic chemotherapy.
* AIDS dementia complex, > or = Stage 2.
* History of zidovudine induced toxicity.
* Any experimental therapy within 30 days.
* Prior history of acute pancreatitis during the past two years or chronic pancreatitis.
* Grade 2 neuropathy.
* Intractable diarrhea.
* History of seizures within the past six months or current requirement of anticonvulsants.
* History of past or current heart disease.
* Fever > 39 C at entry.

Prior Medication:

Excluded:

* Any anti-HIV therapy (other than zidovudine), biologic response modifiers, or pharmacologic doses of corticosteroids within eight weeks of entry (except for the management of severe PCP, in which case duration is not to exceed 21 days).
* Zidovudine therapy for greater than four weeks or prior discontinuation due to drug toxicity.
* Prior therapy with ddI, ddC, D4T, or interferon.
* Any experimental therapy within 30 days.
* Therapy within 30 days with neurotoxic drugs.

Prior Treatment:

Excluded:

* Radiation therapy within two weeks of entry or likely to require radiation therapy (with the exception of electron beam therapy to an area of < 100cm/m2).

Active alcohol or drug abuse, sufficient in the investigator's opinion, to prevent compliance with study therapy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Med Ctr / Main Hosp 4, Washington D.C., District of Columbia
  - Vanderbilt School of Medicine, Nashville, Tennessee
- Saint Vincent's Hosp Med Centre, Darlinghurst, Australia
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico

REFERENCES:
- [Background] Larder BA, Kohli A, Bloor S, Kemp SD, Harrigan PR, Schooley RT, Lange JM, Pennington KN, St Clair MH. Human immunodeficiency virus type 1 drug susceptibility during zidovudine (AZT) monotherapy compared with AZT plus 2',3'-dideoxyinosine or AZT plus 2',3'-dideoxycytidine combination therapy. The protocol 34,225-02 Collaborative Group. J Virol. 1996 Sep;70(9):5922-9. doi: 10.1128/JVI.70.9.5922-5929.1996. PMID 8709213